CLINICAL TRIAL: NCT04760704
Title: Evaluation of the Immunogenicity of mRNA BNT162b2 (COMIRNATY®) Vaccine in Elderly Subjects by Monitoring the Specific Cellular and Humoral Response.
Brief Title: Covid-19 Vaccine Response in Elderly Subjects
Acronym: MONITOCOVAGING
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_02; 2021-A00119-32 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-02-17; First posted 2021-02-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2022-04

CONDITIONS: Covid19 Vaccine
Keywords: SARS-CoV-2; vaccination; immunosenescence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum blood collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Persons aged 65 and over, residing in an institution for dependant elderly or in a long-term care unit
  Interventions: Biological: Specific antibody and cellular immune response after anti-SARS-CoV-2 vaccine administration
- control group: Health and medico-social professionals between 40 and 65 years of age
  Interventions: Biological: Specific antibody and cellular immune response after anti-SARS-CoV-2 vaccine administration

INTERVENTIONS:
Biological: Specific antibody and cellular immune response after anti-SARS-CoV-2 vaccine administration — Specific T cells and specific antibodies assessment

SUMMARY:
The objective of this research is to assess the amplitude and quality of the vaccine response against SARS-CoV-2, defined here by its characteristics established at 3 months, and its persistence over time, defined here at 9 months, in subjects residing in medical establishment for dependent elderly persons, compared to immunocompetent subjects aged 40 to 65 years (control subjects for vaccination over the same period).

ELIGIBILITY:
Inclusion Criteria:

Target population.

* Elderly persons > 65 years old residing in an institution for the elderly or in a long-term care unit for whom an anti-SARS-CoV-2 vaccination is indicated as recommended by French Health Authority (HAS)
* Male or female resident in an institution for the elderly or in a long-term care unit
* For whom consent has been obtained prior to any SARS-CoV-2 vaccination (or from the legal guardian/curator) by COMIRNATY®.
* Having consented to participate in the study, and willing to comply with all study procedures and its duration
* Socially insured patient

Control population

* Health and medico-social sector professionals aged between 40 and 65 years old for whom a COMIRNATY® anti-SARS-CoV-2 vaccination is indicated as recommended by the HAS.
* Male or female between 40 and 65 years of age included
* For whom consent has been obtained prior to any COMIRNATY® SARS-CoV-2 vaccination.
* Having consented to participate in the study, and willing to comply with all study procedures and its duration
* Socially insured subject

Exclusion Criteria, for both groups :

* Progressive infectious pathology
* Progressive neoplastic pathology (or remission of < 5 years)
* Treatment with long-term corticosteroids or immunosuppressants
* Refuse of consent to vaccination or study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly persons > 65 years of age residing in an institution for the elderly or in a long-term care unit for whom an anti-SARS-CoV-2 vaccination is indicated as recommended by French Health Authority (HAS)
Sampling Method: Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Comparison of specific cellular response after anti-SARS-CoV-2 BNT162b2 mRNA vaccine | At 3 months after the first vaccine administration
  Number of gamma interferon-producing anti-S specific T cells detected 3 months after the first vaccine administration between elderly and control subjects

SECONDARY OUTCOMES:
Specific CD4+ and CD8+ T cell response | At 3 months and at 9 months after vaccine administration
  Comparison of number of anti-S specific CD4+ and CD8+ T cells detected at 3 and 9 months, between elderly and control subjects
Total anti-S and neutralizing antibody levels | At 3 months and at 9 months after vaccine administration
  Comparison of total anti-S and neutralizing antibody levels (to pseudo-viral particles and to live virus) at 3 and 9 months after vaccine administration between elderly and control subjects.
Specific immune response according to presence/absence of pre-vaccine antibodies | At 3 months and at 9 months after vaccine administration
  Comparison of anti-S specific T cells, anti-S total antibody and neutralising antibody levels at 3 and 9 months depending on the presence or absence of pre-vaccine antibodies compatible with previous infection in elderly subjects
Specific immune response after COVID-19 vs after BNT162b2 mRNA vaccine | At 3 months after vaccine administration
  Comparison of anti-S-specific total T-cell count, anti-S total antibody levels and neutralising antibody levels 3 months after COVID-19 infection (before any vaccination) and 3 months after vaccination (in subjects who had no COVID-19 before) in elderly subjects
Specific immune response according to nutritional status | At 3 months and at 9 months after vaccine administration
  Correlation between number of anti-S specific T cells, total anti-S antibody and neutralising antibody levels at 3 and 9 months and nutritional status of elderly subjects evaluated according to the Geriatric Nutritional Risk Index (GNRI) in elderly subjects.
Correlation between number of T cells, total anti-S antibody and neutralising antibody at 3 and 9 months, and basal levels of proinflammatory cytokines (interleukin-6, TNF-alpha) in elderly subjects | At 3 months and at 9 months after vaccine administration
Peripheral blood mononuclear cells and serum collection | before the first vaccine injection, 21 days after the first vaccine administration (recall), 28 days after recall, at 3, 6, 9, 12 and 24 months.
  Sampling and conservation of mononuclear cells and serum before injection, at D21 (recall), 28 days after recall, at 3, 6, 9, 12 and 24 months, in elderly and control subjects.
Correlation between number of T cell , total anti-S and neutralizing antibody levels at 3 and 6 months after diagnosis (neutralization tests will be performed on the variant of interest at the time of analysis) | at 3 and 6 months after diagnosis (neutralization tests will be performed on the variant of interest at the time of analysis)
  The neutralizing antibody level at 3 and 6 months will be compared to the levels observed during the infection (serologies done systematically, serum available for retro analysis)
Correlation between number of T-cell , total anti-S and neutralizing antibody levels before the booster and 3, 6 and 12 months after the booster (neutralization tests will be done on BA.1 and any variant of interest at the time of testing). | Before the booster and 3, 6 and 12 months after the booster
Correlation between number of T-cell counts, total anti-S and neutralizing antibody levels within 24-48 hours of a positive PCR (neutralization tests will be done on the variant of interest at the time of testing). | within 24-48 hours of a positive PCR
Saliva samples | at the time of a COVID-19 diagnosis and 3 months after diagnosis, before vaccination or 3, 6 and 12 months after booster.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LEFEVRE, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU lille, Lille, France